CLINICAL TRIAL: NCT07362225
Title: The MPN PROGRESSion Registry: A Retrospective and Prospective Observational Study Collecting Patient-Reported Outcomes, Electronic Health Records, and Claims Data to Track Symptoms, Treatments, and Disease Progression in Individuals Diagnosed With Myeloproliferative Neoplasms (MPNs).
Brief Title: MPN PROGRESSion Registry: Observational Study Tracking Symptoms, Treatments, and Disease Progression in People With Myeloproliferative Neoplasms (MPNs)
Status: Recruiting | Type: Observational
Sponsor: MPN Research Foundation (Other)
Collaborators: Sobi, Inc. (Industry); Karyopharm Therapeutics Inc (Industry); GlaxoSmithKline (Industry); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: MPNRF-PROG-2025-001
Record Dates: First submitted 2026-01-06; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Polycythemia Vera; ET (Essential Thrombocythemia); Polycythemia Vera (PV); Essential Thrombocythemia (ET); Primary Myelofibrosis (MF); Primary Myelofibrosis (PMF); Myelofibrosis; Myelofibrosis (MF); Myelofibrosis, Primary; Myelofibrosis, Post ET; Myelofibrosis, Post PV; Myelofibrosis (PMF); Myelofibrosis，MF; Myelofibrosis; Primary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis; Myelofibrosis Due to and Following Polycythemia Vera; Myelofibrosis Transformation in Essential Thrombocythemia; Myelofibrosis With High Molecular Risk Mutations; MF; Secondary Myelofibrosis; Secondary Myelofibrosis in Myeloproliferative Disease; Secondary Myelofibrosis (Post-Polycythemia Vera Myelofibrosis, Post-Essential Thrombocythemia Myelofibrosis); Post-Polycythemia Vera Myelofibrosis; Post-polycythemia Vera Myelofibrosis (PPV-MF); Post-polycythemia Vera Myelofibrosis (Post-PV MF); Post-polycythemia Vera Myelofibrosis(Post-PV MF); Post-PV MF; Post-Essential Thrombocythemia Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis (PET-MF); Post-essential Thrombocythemia Myelofibrosis(Post-ET MF); Post-essential Thrombocythemia Myelofibrosis (Post-ET MF); Post-ET MF; Pre-fibrotic Myelofibrosis; Myeloproliferative Disorder; Myeloproliferative Disorders; Myeloproliferative Disorders (MPD); Myeloproliferative Neoplasms (MPNs); Myeloproliferative Neoplasm(MPN)-Associated Myelofibrosis; Myeloproliferative Neoplasm With 10% Blasts or Higher; Myeloproliferative Neoplasms; MPN; MPN (Myeloproliferative Neoplasms); MPN-associated Myelofibrosis; Myeloproliferative Neoplasm, Unclassifiable; Myeloproliferative Neoplasm, Not Otherwise Specified; Accelerated Phase MPN; Accelerated Phase Myeloproliferative Neoplasm; Blast Phase MPN; Blast Phase Myeloproliferative Neoplasm; Thrombocythemia Myelofibrosis (PET-MF); Thrombocythemia, Essential; Thrombocythemia, Hemorrhagic; Agnogenic Myeloid Metaplasia; Chronic Idiopathic Myelofibrosis; Idiopathic Myelofibrosis; MDS/MPN Crossover Syndromes
Keywords: Myeloproliferative Neoplasms; Polycythemia Vera; Essential Thrombocythemia; Secondary Myelofibrosis; Pre-fibrotic Primary Myelofibrosis; Myeloproliferative Disorder; Myeloproliferative Neoplasm, Unclassifiable; Myeloproliferative Neoplasm, Accelerated Phase; Myeloproliferative Neoplasm, Blast Phase; Chronic Myeloproliferative Disease; Hematologic Neoplasms; Bone Marrow Neoplasms; Blood Cancer; Disease Progression; Biomarker Discovery; Patient-Reported Outcomes; Electronic Health Records; Real-World Evidence; Longitudinal Study; Observational Study; Registry Study; Natural History Study; Quality of Life; Rare Diseases; Chronic Hematologic Diseases; Risk Stratification; Symptom Burden; Medical Claims Data; Longitudinal Data Collection; Patient-Centered Research; Health Outcomes Research; Clinical Outcomes; Clinical Guidelines Development; Regulatory Science; Drug Development; Treatment Response
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis; Myeloproliferative Disorders; Blast Crisis; Hematologic Neoplasms; Bone Marrow Neoplasms; Disease Progression; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MPN Patient Cohort: Adults (18 years and older) diagnosed with a myeloproliferative neoplasm (MPN), including polycythemia vera (PV), essential thrombocythemia (ET), primary myelofibrosis (MF), secondary myelofibrosis, pre-fibrotic primary myelofibrosis (pre-PMF), myeloproliferative neoplasm-unclassifiable (MPN-U), myeloproliferative neoplasm-accelerated phase (MPN-AP), myeloproliferative neoplasm-blast phase (MPN-BP), or post-MPN acute myeloid leukemia (AML), and myelodysplastic syndrome (MDS)/MPN overlap syndrome as defined above per WHO 2022 criteria, including patients originally diagnosed with one of these conditions but who have received one or more stem cell transplants (SCTs) or bone marrow transplants (BMTs) enrolled in a prospective observational registry study to track clinical outcomes, disease progression, treatment patterns, patient-reported outcomes, and long-term health trajectories over time.

SUMMARY:
The MPN PROGRESSion Registry is a multi-year, observational research study designed to improve understanding of myeloproliferative neoplasms (MPNs)-a group of rare, chronic blood cancers that include polycythemia vera (PV), essential thrombocythemia (ET), primary myelofibrosis (MF), pre-fibrotic primary myelofibrosis (pre-PMF), secondary myelofibrosis, myeloproliferative neoplasm-unclassifiable (MPN-U), MPN in accelerated phase (MPN-AP), and MPN in blast phase (MPN-BP), post-MPN Acute Myeloid Leukemia (AML), and MDS/MPN overlap syndrome as defined above per WHO 2022 criteria, including patients originally diagnosed with one of these conditions but who have received one or more SCTs and/or BMTs . These conditions are characterized by abnormal blood cell production in the bone marrow and may lead to complications such as blood clots, bleeding, bone marrow fibrosis, and, in some cases, progression to acute leukemia.

The central hypothesis of the registry is that collecting and analyzing real-world, longitudinal data-including electronic health records (EHRs), laboratory values, treatments, and patient-reported outcomes (PROs)-from a diverse population of people living with MPNs will help identify patterns and predictors of disease progression, treatment response, quality of life, and long-term outcomes. These insights are intended to guide future research, inform clinical guidelines, and support improvements in patient care.

The registry is non-interventional and observational; participants do not receive investigational treatments, and all medical care continues under the supervision of their own physicians. Data collection includes EHRs, PRO surveys, patient-reported symptom and lab tracking, insurance claims, and, in the future, may include linkages with other relevant disease registries and datasets. Potential collaborations under consideration include those with the European LeukemiaNet (ELN) MPN Registry, the Mayo Clinic MPN Database, the Center for International Blood and Marrow Transplant Research (CIBMTR), the SEER Program, Harmony Alliance Foundation, and the National Cancer Database (NCDB).

The registry emphasizes the patient voice, incorporating lived experiences related to hallmark MPN symptoms such as fatigue, pruritus (itching), bone pain, night sweats, and social and emotional impacts. Participants will be followed for at least five years, with many enrolled for ten years or longer, to capture the natural history of disease and long-term outcomes. PRO surveys will be completed approximately every six months, and EHR data will be regularly reviewed to track changes in clinical status, treatment, and disease evolution.

Statistical analyses will use descriptive and inferential methods to examine clinical characteristics, symptom burden, disease trajectories, and patient-centered outcomes. Planned subgroup analyses may compare differences across diagnoses, treatment approaches, demographics, or genomic factors. Analytic plans will be finalized during the course of the study and may evolve in response to emerging scientific questions.

The registry is open to adults (18 years or older) living in the United States who have been diagnosed with any of the included MPN subtypes and are willing to share health information and complete study surveys. Individuals currently enrolled in interventional clinical trials or unable to provide informed consent may be excluded. Participation is voluntary, and participants may withdraw from the study at any time without affecting their medical care.

Privacy and data security are core priorities. Participant data will be securely stored and managed in accordance with all applicable privacy laws and research regulations. No identifiable information will be shared with external parties without appropriate authorization. Oversight is provided by a Steering Committee and a Patient Engagement Advisory Committee (PEAC), ensuring rigorous scientific, ethical, and patient-centered governance.

The registry is sponsored by the MPN Research Foundation, a nonprofit organization advancing research and patient advocacy in myeloproliferative neoplasms (MPNs). Participants can contact the registry team at any time with questions and will receive periodic updates on study findings.

This study aims to address critical gaps in understanding the real-world experiences of people with MPNs-such as symptom burden over time, risk factors for progression, and how different treatments impact patient outcomes. Findings may inform clinical trial design, support biomarker discovery, and contribute to the development of updated treatment recommendations. The registry is committed to including participants from diverse backgrounds and clinical settings to ensure findings are broadly applicable across the MPN community. Summary results will be shared through scientific publications, presentations, and other dissemination efforts to advance MPN research and care globally.

DETAILED DESCRIPTION:
The MPN PROGRESSion Registry is a U.S.-based, prospective, observational, non-interventional study designed to track long-term clinical outcomes, treatment patterns, symptoms, quality of life, and disease progression in individuals diagnosed with myeloproliferative neoplasms (MPNs). Eligible subtypes include polycythemia vera (PV), essential thrombocythemia (ET), primary myelofibrosis (MF), secondary MF, pre-fibrotic primary myelofibrosis (pre-PMF), myeloproliferative neoplasm-unclassifiable (MPN-U), MPN in accelerated phase (MPN-AP), MDS/MPN Overlap Syndrome, and MPN in blast phase (MPN-BP), as defined by WHO 2022 criteria, including patients originally diagnosed with one of these conditions but who have received one or more stem cell transplant (SCT)s and/or bone marrow transplant (BMT)s.

The registry integrates multimodal data sources-including structured electronic health record (EHR) extractions, patient-reported outcomes (PROs), medical claims, and potential future linkages with external disease registries-to generate a comprehensive, real-world dataset. This approach supports the identification of factors associated with disease trajectory, treatment response, symptom burden, and healthcare utilization, with the goal of advancing observational research, informing clinical care, and supporting regulatory science.

Participants will be enrolled over a minimum of five years, with many expected to remain in the registry for ten years or longer. An initial run-in phase aims to enroll approximately 1,500 participants to assess operational feasibility, data completeness, retention strategies, and analytic approaches. Over time, the registry will expand to include a broader, more diverse cohort capable of supporting subgroup analyses and capturing rare progression events.

The registry emphasizes patient engagement through structured PRO collection and personalized communications. PROs are collected on a tiered schedule to balance participant burden with scientific value. The MPN-SAF Total Symptom Score (TSS) and PGI-S (Patient Global Impression of Severity) are collected every three months to assess symptom burden and global health status. Every six months, participants also complete additional PROs including the EORTC QLQ-C30 (quality of life), an IRB approved Modified-PHQ-9 (mental health), and PROMIS Fatigue 8a. These PROs are supplemented by EHR refreshes, claims data, and mortality data linkages at the same six-month intervals. Participants receive automated reminders, and support is available from patient navigators. Additional engagement includes study updates, webinars, and optional non-monetary incentives.

Governance is provided by a Steering Committee composed of scientific and clinical experts and a Patient Engagement Advisory Committee (PEAC) that includes patients and caregivers from diverse backgrounds. These bodies provide ongoing oversight, ensure patient-centered governance, and advise on scientific, operational, and ethical matters. The study is approved by a central institutional review board (IRB) and complies with Good Clinical Practice (GCP), HIPAA, and all applicable regulatory standards. Participation does not influence medical care, and all treatment decisions remain solely between patients and their healthcare providers.

The registry operates under a formal quality assurance framework that includes automated and manual data validation, internal monitoring, and regular data audits. Range checks, logic rules, and reconciliation of EHR, PRO, and claims data are used to enhance data completeness and accuracy. Data elements are defined through a structured data dictionary that includes descriptions, formats, allowable ranges, and coding systems (e.g., ICD-10, SNOMED CT, LOINC, MedDRA), which is updated as needed through a documented change control process.

Personally identifiable information (PII) is separated from research data using an Honest Broker model, with encryption, access controls, and full audit trails ensuring data security and participant confidentiality. The registry complies with applicable U.S. privacy regulations, and participants may withdraw consent at any time. Data collected prior to withdrawal may continue to be used unless otherwise requested and feasible.

Statistical analyses will apply descriptive and inferential methods to examine clinical characteristics, symptom burden, treatment patterns, and progression events. Planned analyses may include comparisons across diagnostic subtypes, treatment strategies, demographics, or genetic factors. The formal statistical analysis plan (SAP) will be finalized after initial data review and is expected to evolve based on emerging scientific priorities. At this time, no independent data monitoring committee (DMC) is in place.

Planned exploratory analyses may also include comparisons or potential data harmonization with external resources such as the European LeukemiaNet (ELN) MPN Registry, the Mayo Clinic MPN Database, the Center for International Blood and Marrow Transplant Research (CIBMTR), the Surveillance, Epidemiology, and End Results (SEER) Program, the Harmony Alliance Foundation, and the National Cancer Database (NCDB), contingent on future partnerships and data-sharing agreements.

The real-world evidence (RWE) generated by this registry is intended to support a range of research goals, including understanding natural disease history, identifying risk factors, evaluating patient-reported outcomes over time, and informing the development of biomarkers and surrogate endpoints. Findings may help shape future clinical trial design, therapeutic strategies, and policy guidance. Dissemination will occur through peer-reviewed publications, conference presentations, and participant-facing summaries to ensure transparency and impact across the broader MPN community.

The registry is sponsored and administered by the MPN Research Foundation, a nonprofit organization advancing research and patient advocacy in myeloproliferative neoplasms (MPNs).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older at the time of enrollment.
* Confirmed diagnosis of a myeloproliferative neoplasm (MPN), including one or more of the following subtypes, according to WHO 2022 criteria, including patients originally diagnosed with one of these conditions but who have received one or more stem cell transplants (SCTs) or bone marrow transplants (BMTs):
* Polycythemia vera (PV)
* Essential thrombocythemia (ET)
* Primary myelofibrosis (PMF)
* Secondary myelofibrosis (post-ET or post-PV MF)
* Pre-fibrotic primary myelofibrosis (pre-PMF)
* Myeloproliferative neoplasm-unclassifiable (MPN-U)
* Myeloproliferative neoplasm, accelerated phase (MPN-AP)
* Myeloproliferative neoplasm, blast phase (MPN-BP)
* Post-MPN acute myeloid leukemia (AML)
* Myelodysplastic syndrome (MDS)/MPN overlap syndrome
* Myeloproliferative neoplasm, blast phase (MPN-BP)
* Ability to provide informed consent electronically or through a legally authorized representative.
* Willingness to share health information, including electronic health records (EHR), laboratory values, and survey responses.
* Willingness to complete periodic patient-reported outcome (PRO) surveys and symptom tracking assessments.

Exclusion Criteria:

* Individuals under 18 years of age.
* Inability to provide informed consent, either directly or through a legally authorized representative.
* Currently enrolled in an interventional clinical trial where participation would interfere with the ability to participate in this observational registry (based on investigator or sponsor judgment).
* Any condition that, in the judgment of the study team, would make participation in the registry infeasible or unsafe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18 years and older) diagnosed with a myeloproliferative neoplasm (MPN), including polycythemia vera, essential thrombocythemia, primary myelofibrosis, secondary myelofibrosis, pre-fibrotic primary myelofibrosis, MPN-unclassifiable, MPN-accelerated phase, or MPN-blast phase, post-MPN AML, or MDS/MPN overlap syndrome (including patients originally diagnosed with one of these conditions but who have received one or more SCTs or BMTs) residing in the United States. Participants are enrolled exclusively through direct-to-patient outreach using online recruitment, social media, digital advertising, and patient advocacy networks. All participants must provide electronic informed consent, have accessible electronic health record (EHR) data, and be willing to complete digital patient-reported outcome surveys. The study aims to capture a diverse national cohort for real-world, longitudinal research on disease progression, treatment patterns, and outcomes .
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2035-09-08 (Estimated); Study Completion 2035-09-08 (Estimated)

PRIMARY OUTCOMES:
Time to Disease Progression | Assessed continuously from enrollment over a minimum of 5 years per participant, with extended follow-up beyond 10 years for participants who remain active in the registry.
  Time from enrollment to the first documented disease progression event, defined as transformation between MPN subtypes (for example, essential thrombocythemia or polycythemia vera to myelofibrosis), development of accelerated-phase MPN (MPN-AP), progression to blast phase (MPN-BP), or meeting updated World Health Organization (WHO) or International Working Group for Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) criteria for disease progression. This outcome measures the rate and timing of disease evolution over time and evaluates associations with treatments, exposures, and clinical risk factors among adults diagnosed with MPNs.

SECONDARY OUTCOMES:
Overall Survival | Assessed continuously from enrollment over a minimum of 5 years per participant, with extended follow-up beyond 10 years for active participants.
  Time from enrollment to death from any cause among participants diagnosed with an MPN. This outcome measures overall survival patterns and examines associations between survival and treatments, risk factors, exposures, and clinical characteristics over time.
Change in MPN-SAF Total Symptom Score (TSS) | Assessed every 3-6 months over a minimum of 5 years per participant, with extended follow-up beyond 10 years where applicable.
  The MPN-SAF TSS patient reported outcome (PRO) tool tracks MPN symptoms, including fatigue, pruritus, night sweats, bone pain, and early satiety.
Event-Free Survival | Assessed continuously from enrollment over a minimum of 5 years per participant, with extended follow-up beyond 10 years where applicable.
  Time from enrollment to first occurrence of a progression event, transformation to accelerated or blast phase, or death from any cause. This outcome provides an integrated measure of survival and disease stability among participants diagnosed with MPNs.
Patient Global Impression Scale - Severity (PGI-S) | Time Frame: Assessed every 3-6 months over a minimum of 5 years per participant, with extended follow-up beyond 10 years where applicable.
  The PGI-S is a PRO that captures patient-perceived overall change in health status over time.
EORTC QLG Core Questionnaire (QLQ-C30 | Time Frame: Assessed every 3-6 months over a minimum of 5 years per participant, with extended follow-up beyond 10 years where applicable.
  The EORTC QLQ-C30 is a 30 item PRO that evaluates overall health-related quality of life, including functional status and symptom burden.
Modified Patient Health Questionnaire (PHQ-9) | Time Frame: Assessed every 3-6 months over a minimum of 5 years per participant, with extended follow-up beyond 10 years where applicable.
  The Modified PHQ-9 is a PRO that screens for depressive symptoms commonly observed in MPN patients.
Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Fatigue 8a: Assesses fatigue in MPN patients, specifically targeting the experience of fatigue and its impact on daily life. | Time Frame: Assessed every 3-6 months over a minimum of 5 years per participant, with extended follow-up beyond 10 years where applicable.
  The PROMIS Short Form v1.0 - Fatigue 8a is a PRO that assesses fatigue in MPN patients, specifically targeting the experience of fatigue and its impact on daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Raajit Rampal, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - MPN Research Foundation, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No
The MPN PROGRESSion Registry does not plan to share individual participant data (IPD) outside the study team, sponsor, and designated governance committees. Due to the sensitive nature of patient health data and the direct-to-patient enrollment model, sharing of IPD is restricted to protect participant privacy and comply with applicable privacy laws, ethical standards, and institutional review board (IRB) requirements. Aggregate, de-identified results may be shared through scientific publications, conference presentations, and summary reports, but no participant-level data will be made publicly available.

REFERENCES:
- See also: MPN Research Foundation MPN PROGRESSion Registry Webpage — https://mpnresearchfoundation.org/mpnprogressionregistry/

DOCUMENTS (2):
  • Study Protocol (2025-11-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT07362225/Prot_000.pdf
  • Informed Consent Form (2025-11-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT07362225/ICF_001.pdf